CLINICAL TRIAL: NCT00665444
Title: Reducing Medical Risks in Individuals With Bipolar Disorder: Enhancing Outcomes With Aripiprazole
Brief Title: Study of Aripiprazole to Reduce Medical Risks in Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated by the sponser due to low study enrollment.
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Holly Swartz, Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMS.WPIC.I#0008449
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Bipolar Disorder; Metabolic Syndrome
Keywords: bipolar disorder; sedation; overweight; Abilify; medication
MeSH Terms: conditions — Bipolar Disorder; Metabolic Syndrome; Overweight | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Aripiprazole
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — All subjects will be assessed at baseline and then switched from their current antimanic agent to aripiprazole. Arpipirazole will be titrated from a starting dose of 5 mg/day up to a target dose of 15 mg/day over a period of up to 2 months (approximately 8 weeks). Concomitant medication will not be changed unless medically necessary. If a subject is taking an antipsychotic in addition to divalproex, aripiprazole will replace the antipsychotic.
  Other Names: Abilify

SUMMARY:
The proposed study is a non-randomized, open label trial that will examine the potential to reduce metabolic risk factors in patients with bipolar I disorder and improve psychiatric and functional outcomes. To accomplish our objective, we plan to conduct a 5-month intervention of 50 obese or overweight adults diagnosed with bipolar disorder. The study will be divided in three steps: Screening, Baseline Period (cross taper to aripiprazole, up to 2 months in duration), Months 1-3 (continued aripiprazole treatment). Subjects will be assessed and meet with their study psychiatrist at least bi-monthly throughout their participation, more frequently when clinically necessary (e.g. during medication tapering or if manic/depressive symptoms emerge). Brief clinical assessments will be conducted at each visit. More thorough assessments will be conducted at Baseline, Week 2, and Month 3.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Body mass index (BMI) >=25;
3. Currently taking a regimen of medications for bipolar disorder likely to cause, sedation, weight gain or undesirable metabolic effects;
4. Able to give basic informed consent
5. Meets DSM-IV criteria for lifetime bipolar I or II disorder and are presently in sustained remission (CGI BP<3 in the previous 8-week period measured through a complete psychiatric history at screening and patient report.)
6. Epworth Scale Score > 7
7. Women of childbearing potential must agree to use a doctor-approved birth control throughout participation in the study

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements (i.e., complete forms, attend scheduled evaluations)
2. Not competent to provide informed consent in the opinion of the investigator
3. Ultra-rapid cycling (>4 episodes per month) bipolar I disorder
4. Unstable and severe medical illness that requires immediate and intensive medical attention, When appropriate, the patients can be reconsidered for inclusion in the study if/when their medical condition becomes compatible with participation in a protocol-driven research study
5. Women who are planning to become pregnant, currently pregnant, or breast-feeding;
6. Current substance dependence; however, if a subject only has substance abuse/use, after the first positive drug screen, another drug screen will be repeated. If that drug screen is positive, the subject will be excluded. If the second drug screen is negative, the subject will be considered for the study;
7. Subjects who have previously failed an adequate trial of aripiprazole.
8. Subjects with a suicide attempt in the past 2 years;
9. Subjects with a history of inpatient admission in the past 1 year;
10. Subjects with a history of homicidal ideation;
11. Any subject for whom the PI deems that the potential risks in participating in the study outweigh the potential benefits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Aripiprazole
  Aripiprazole: All subjects will be assessed at baseline and then switched from their current antimanic agent to aripiprazole. Arpipirazole will be titrated from a starting dose of 5 mg/day up to a target dose of 15 mg/day over a period of up to 2 months (approximately 8 weeks). Concomitant medication will not be changed unless medically necessary. If a subject is taking an antipsychotic in addition to divalproex, aripiprazole will replace the antipsychotic.
Period: Overall Study
Arm/Group | Aripiprazole
Started | 3
Completed | 1
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Study Terminated by Study Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: BodyMedia Armband (Sleep/Wake and Activity/Inactivity Patterns),
Time Frame: 3 months
Population: 0-the study was terminated early by the study sponsor due to low enrollment numbers. Only one participant completed the study in its duration and the study was terminated before any outcome data could be analyzed.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

2. Primary Outcome: Epworth Sleepiness Scale (General Level of Daytime Sleepiness)
Time Frame: 3 month
Population: as for outcome 1
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

3. Secondary Outcome: Global Assessment of Functioning
Time Frame: 3 months
Population: Study was terminated early and data were not collected for this outcome.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life Enjoyment Questionnaire
Time Frame: 3 months
Population: Study was terminated early and data were not collected for this outcome.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

5. Secondary Outcome: Young Mania Rating Scale
Time Frame: 3 months
Population: Study was terminated early and data were not collected for this outcome.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

6. Secondary Outcome: Hamilton Rating Scale for Depression
Time Frame: 3 months
Population: Study was terminated early and data were not collected for this outcome.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
the study was terminated early by the study sponsor due to low enrol...

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No